CLINICAL TRIAL: NCT00817219
Title: Safety and Efficacy of TACLONEX Ointment in Adolescent Patients (Aged 12 to 17 Years) With Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCB 0501 INT
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Results first posted 2013-01-07 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2015-03

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TACLONEX ointment (Experimental)
  Interventions: Drug: Calcipotriene plus betamethasone dipropionate ointment

INTERVENTIONS:
Drug: Calcipotriene plus betamethasone dipropionate ointment — Once daily application for 4 weeks

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of 4 weeks of TACLONEX ointment in adolescent patients with psoriasis vulgaris.

DETAILED DESCRIPTION:
TACLONEX ointment has marketing approval in many countries for the treatment of psoriasis vulgaris in adults. No studies have been conducted in patients less than 18 years of age. However, about 25% of affected individuals are diagnosed between 10 and 19 years of age, hence psoriasis is also prevalent in the adolescent age group (12-17 years).

All patients will receive TACLONEX. To evaluate the safety of TACLONEX ointment, all adverse events will be recorded. In addition, any systemic absorption of the active components, betamethasone dipropionate and calcipotriene, will be evaluated by assessing adrenal function (using CORTROSYN™ test) and calcium metabolism (by measuring serum calcium and the urinary calcium:creatinine ratio), respectively.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 to 17 years, inclusive.
* Psoriasis vulgaris on the trunk and/or limbs which is:
* amenable to topical treatment
* of an extent of 5-30% of BSA
* of at least a moderate severity
* A serum cortisol concentration above 5 mcg/dL before ACTH-challenge and above 18 mcg/dL at 30 minutes after ACTH-challenge.
* Albumin-corrected serum calcium and urinary calcium:creatinine ratio within the reference range.

Exclusion Criteria:

* Serious allergy, serious asthma, or serious allergic skin rash.
* A history of sensitivity to any medication.
* PUVA or Grenz ray therapy, UVB therapy, systemic treatment with biological therapies, corticosteroids, or other therapies with an effect on psoriasis, topical treatment with corticosteroids or vitamin D analogues, treatment with enzymatic inductors, cytochrome P450 inhibitors, hypoglycemic sulfonamides, antidepressive medications, estrogen therapy, calcium supplements or vitamin D supplements.
* Guttate, erythrodermic, exfoliative or pustular psoriasis.
* Viral lesions of the skin, fungal or bacterial skin infections, ulcers or wounds.
* Severe renal insufficiency, severe hepatic disorders, disorders of calcium metabolism associated with hypercalcemia, any cardiac condition or endocrine disorder.
* Diabetes mellitus
* Cushing's disease or Addison's disease.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy S Paller, MD, Principal Investigator — Northwestern University's Feinberg School of Medicine
Locations (8):
- United States (8):
  - Center for Dermatology Clinical Research, Fremont, California
  - University of California at San Diego/Rady Children's Hospital, San Diego, California
  - Ameriderm Research, Maitland, Florida
  - Northwestern University's Feinberg School of Medicine, Chicago, Illinois
  - Arlington Research Center, Arlington, Texas
  - University of Texas-Dermatology, Houston, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - DBA Dermatology Associates, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study period was 15 July 2009 (date of first subject's first screening visit) to 05 December 2011 (date of the last subject's last on-treatment visit)
Pre-assignment Details: Before starting treatment there was a washout/screening phase lasting for 3 days to 6 weeks, depending on the prior use of excluded treatments.
Groups:
- TACLONEX Ointment: TACLONEX (Calcipotriol and betamethasone dipropionate) ointment applied once daily to psoriasis on the trunk/limbs for 4 weeks
Period: Overall Study
Arm/Group | TACLONEX Ointment
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TACLONEX Ointment
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Adverse Drug Reactions
Description: The number of participants experiencing each type of adverse drug reaction. Adverse drug reactions were defined as adverse events for which the investigator had not described the causal relationship to trial medication as "not related".
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | TACLONEX Ointment
Number analyzed (Participants) | 33
participants | 2

2. Primary Outcome: Serum Cortisol Concentration of ≤18 mcg/dL at 30 Minutes After ACTH-challenge at End of Treatment
Description: The ACTH(Adrenocorticotropic hormone)-challenge test involves injecting a synthetic subunit of ACTH into the patient,and measuring the cortisol produced by the adrenal glands 30 and 60 minutes after the injection.
Time Frame: Week 4
Population: One participant did not provide data for the ACTH-challenge test following the start of treatment, thus only 32 participants were included in this analysis
Measure: Number; unit: participants
Arm/Group | TACLONEX Ointment
Number analyzed (Participants) | 32
participants | 0

3. Primary Outcome: Serum Cortisol Concentration of ≤18 mcg/dL at 30 and 60 Minutes After ACTH-challenge at End of Treatment
Description: as for outcome 2
Time Frame: Week 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | TACLONEX Ointment
Number analyzed (Participants) | 32
participants | 0

4. Primary Outcome: Change in Albumin Corrected Serum Calcium From Baseline to End of Treatment
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | TACLONEX Ointment
Number analyzed (Participants) | 33
mmol/L | 0.005 (0.094)

5. Primary Outcome: Change in Urinary Calcium:Creatinine Ratio From Baseline to End of Treatment.
Time Frame: Baseline and 4 Weeks
Measure: Mean (Standard Deviation); unit: mmol/g
Arm/Group | TACLONEX Ointment
Number analyzed (Participants) | 33
mmol/g | 0.717 (2.877)

6. Secondary Outcome: "Controlled Disease"(i.e., "Clear" or "Almost Clear") According to the Investigator's Global Assessment of Disease Severity at Week 4.
Description: The investigator made an assessment of the disease severity (Plaque thickening, Scaling and Erythema) using a 6-point scale (Clear, Almost clear, Mild, Moderate, Severe, and Very severe). This assessment represented the average lesion severity on the trunk and limbs.
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | TACLONEX Ointment
Number analyzed (Participants) | 33
participants | 20

7. Secondary Outcome: "Controlled Disease"(i.e., "Clear" or "Very Mild") According to the Patient's Global Assessment of Disease Severity at Week 4.
Description: The patient made an assessment of the disease severity using a 5-point scale (Clear, Very Mild, Mild, Moderate, and Severe).
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | TACLONEX Ointment
Number analyzed (Participants) | 33
participants | 23

8. Secondary Outcome: Percentage Change in PASI From Baseline to Week 4.
Description: PASI is Psoriasis Area and Severity Index and is based on the investigator's assessment of extent and severity of the disease. It can range from 0 (best) to 64.8(worst). The PASI used in this trial is modified to exclude assessment of the head, as trial treatment is not used here.
Time Frame: Baseline and 4 weeks
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | TACLONEX Ointment
Number analyzed (Participants) | 33
percentage | -72.5 [-81.1 to -63.9]

9. Secondary Outcome: PASI 75 at Week 4.
Description: PASI 75 is at least 75% reduction in PASI from baseline. PASI is Psoriasis Area and Severity Index and is based on the investigator's assessment of extent and severity of the disease. It can range from 0 (best) to 64.8(worst). The PASI used in this trial is modified to exclude assessment of the head, as trial treatment is not used here.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | TACLONEX Ointment
Number analyzed (Participants) | 33
participants | 17

10. Secondary Outcome: PASI 50 at Week 4.
Description: PASI 50 is at least 50% reduction in PASI from baseline. PASI is Psoriasis Area and Severity Index and is based on the investigator'sassessment of extent and severity of the disease. It can range from 0 (best) to 64.8(worst). The PASI used in this trial is modified to exclude assessment of the head, as trial treatment is not used here.
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | TACLONEX Ointment
Number analyzed (Participants) | 33
participants | 28

ADVERSE EVENTS:
Arm/Group | TACLONEX Ointment
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 10/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TACLONEX Ointment (N=33)
Upper respiratory tract (Infections and infestations) | 2
Headache (Nervous system disorders) | 2
Tension headache (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Rash papular (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review at least 30 days prior to the same paper being submitted for publication or presentation. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.